CLINICAL TRIAL: NCT05265780
Title: Effect of Kinesiotaping on Elbow Joint Proprioception
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Dokuz Eylul University (Other)
Responsible Party: Principal Investigator, Kevser Sevik, Principal Investigator, Dokuz Eylul University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: DokuzEU131314
Record Dates: First submitted 2022-02-17; First posted 2022-03-04 (Actual); Last update posted 2022-03-04 (Actual); Status verified 2022-03

CONDITIONS: Healthy
MeSH Terms: interventions — Athletic Tape

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- kinesiotape (Experimental): kinesiotaping group
  Interventions: Procedure: kinesiotape
- control (Sham Comparator): sham group
  Interventions: Procedure: sham taping

INTERVENTIONS:
Procedure: kinesiotape — an elastic adhesive tape
  Arms: kinesiotape
Procedure: sham taping — a sham taping without the tension
  Arms: control

SUMMARY:
assessing the effects of kinesiotape application on elbow joint proprioception

DETAILED DESCRIPTION:
assessing the effects of kinesiotape application on elbow joint proprioception by evaluating joint position sense

ELIGIBILITY:
Inclusion Criteria:

* 18-85 years

Exclusion Criteria:

* any elbow disorders
* any neurological disorders

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 48 (Actual)
Dates: Start 2021-10-01 (Actual); Primary Completion 2021-12-01 (Actual); Study Completion 2022-01-01 (Actual)

PRIMARY OUTCOMES:
proprioception by evaluating the joint position sense | 35 minutes
  proprioception by evaluating the joint position sense of the elbow at 70 and 100 degrees of flexion

CONTACTS AND LOCATIONS:
Overall Officials: kevser sevik, Principal Investigator — Dokuz Eylul University
Locations (1):
- School of Physical Therapy and Rehabilitation, Balçova, İzmir, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No